CLINICAL TRIAL: NCT00776568
Title: Extracorporeal Shock Wave Therapy (ESWT) for the Treatment of Refractory Angina Pectoris
Brief Title: Treatment of Refractory Angina Pectoris by Shock Wave Therapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universal Research Group (Network)
Collaborators: UNIQUIP INTERNATIONAL, Pakistan (Unknown)
Responsible Party: Executive Director, Karachi Institute of Heart Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URG/UQ/002/01; ISRCTN68966125
Record Dates: First submitted 2008-10-20; First posted 2008-10-21 (Estimated); Last update posted 2008-10-21 (Estimated); Status verified 2008-10

CONDITIONS: Angina Pectoris
MeSH Terms: conditions — Angina Pectoris | interventions — Antihypertensive Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Active Comparator)
  Interventions: Drug: Anti-hypertensive drugs
- 1 (Experimental)
  Interventions: Procedure: Extra-corporeal shockwave

INTERVENTIONS:
Procedure: Extra-corporeal shockwave — Low intensity shock waves are applied as 300 shocks per visit for 09 visits. The treatment visit is carried at week 1, 5 and 9.
  Arms: 1
Drug: Anti-hypertensive drugs — ACE inhibitors, Ca channel blockers, Beta blockers, Diuretics, Cholesterol lowering agents and/or other drugs used alone or in combination, as prescribed.
  Arms: 2

SUMMARY:
The purpose of this study is to determine that extracorporeal shock wave therapy (ESWT) is safe and effective for the treatment of refractory angina pectoris.

DETAILED DESCRIPTION:
Patients with advanced CAD frequently have limited symptoms with recurrent angina, angina at low work thresholds, breathlessness, and other debilitating conditions. These patients have often been through several "re-do" coronary bypass procedures and multiple percutaneous coronary interventions.

Surgical and interventional options for these patients typically have been exhausted or will result in only partial revascularization. Therefore, therapy remains limited to the use of multiple anti-anginal medications, reduced activity, exertion, and stress level, and significant alteration and limitation of lifestyle.

The goal of this emerging approach is to therapeutically induce the growth and development of new vasculature in zones of severe ischemia in the myocardium, with the hope that new capillaries and arterioles generated will connect to remnant existing vasculature. These neovessels are viewed to act as collaterals, perfusing ischemic territories unapproachable by macro procedures such as PCI and/or CABG.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years or older.
* Diagnosis of chronic stable angina pectoris. Diagnosis is based on medical history, complete physical evaluation, and Exercise Single-Photon Emission Computed Tomography (Exercise SPECT).
* Patient has documented myocardial segments with reversible ischemia and or hibernation.
* Patient is classified as AP CCS of III or IV.
* Patient should be on a stable dosage of medication used to treat angina for at least 6 weeks prior to enrollment.
* Patients demonstrates exercise tolerance time (ETT) duration <10 minutes on a modified Bruce protocol on 2 consecutive tests (tests no less than 24 hours and no more than 2 weeks apart), with the second test within 25% of the first (Patients should not be informed of exercise restrictions required for entry into the study).
* Patient has refused to undergo another angioplasty or CABG.
* Patient has signed an informed consent form.
* Patient's condition should be stable and should have a life expectancy of >12 months.
* Patient's current and past medical condition and status will be assessed using previous medical history, physical evaluation, and the physicians (principle investigator's) medical opinion.
* Newly diagnosed type II diabetes.

Exclusion Criteria:

* Chronic lung disease including emphysema and pulmonary fibrosis.
* Active endocarditis, myocarditis or pericarditis.
* Patient is simultaneously participating in another device or drug study, or has participated in any
* Clinical trial involving an experimental device or drug, including other drugs or devices enhancing cardiac neovascularization, or any ESWT machine for neovascularization of a competitor company within 3 months of entry into the study.
* Patients who are unwilling or unable to cooperate with study procedure.
* Patients who are unwilling to quit smoking during the study procedure (including screening phase)
* Patients who had myocardial infarction (MI) less than 3 months prior to treatment.
* Patients who are diagnosed with a 3rd and 4th degree heart valve disease.
* Patient with intraventricular thrombus.
* Pregnancy.
* Patient with a malignancy in the area of treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-02; Primary Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
Alleviation of anginal symptoms | 06 months

SECONDARY OUTCOMES:
The change in SPECT in perfusion from baseline to 6 months post-baseline (17 segments model | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Abdul Samad, MD, Principal Investigator — Karachi Institute of Heart Diseases
Locations (1):
- Karachi Institute of Heart Diseases, Karachi, Pakistan

REFERENCES:
- See also: Related Info — http://www.controlled-trials.com/ISRCTN68966125